CLINICAL TRIAL: NCT05632055
Title: miRNA and FGF21 Profile in First Trimester and Efficacy of Gestational Diabetes Prediction and Pregnancy Outcomes
Brief Title: miRNA (microRNA) and FGF21 (Fibroblast Growth Factor-21) Profile in First Trimester and Gestational Diabetes Prediction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kuntharee Traisrisilp, Associate Professor, Chiang Mai University
Other Study IDs: OBG-2563-07494
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancy with GDM: Pregnant women who positive test for 100gm OGTT (abnormal 2 or more blood glucose level according NDDG (National Diabetes Data Group) criteria)
  Interventions: Other: blood draw
- Pregnancy without GDM: Pregnant women who negative test for 100gm OGTT
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Blood test for miRNA and FGF21. However, the laboratory result is not reported and not involved in management

SUMMARY:
The goal of this observational study is to compare miRNA and FGF21 in pregnancy with and without GDM (Gestational Diabetes) The main question it aims to answer that miRNA and FGF21 are different between two groups.

Participants will be retrieved blood sample during first trimester and undergone 100 gm OGTT (oral glucose challenge test) during 24-28 weeks of gestation.

DETAILED DESCRIPTION:
Pregnant women who attended antenatal care at Maharaj Nakorn Chiang Mai hospital during first trimester were recruited.

Participants received routine standard prenatal care except,

1. additional blood test during 11-13 week 6 days (Blood was collected for further analysis)
2. performed 75gm OGTT during 24-28 week

Baseline data and pregnancy outcome were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women who attend at our clinic in first trimester

Exclusion Criteria:

* known underlying disease such as chronic hypertension, pregestational diabetes, SLE
* normal structural fetal anatomical screening
* incomplete obstetric data

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — because we study in pregnancy woman
Study Population: Healthy pregnant women with single alive fetus Participants will be subgroup based on the result of 100gm OGTT
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2000-08-26 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
miRNA profile | within 1 month after blood drawn
  miRNA profile in first trimester of pregnancy and efficacy for GDM prediction

SECONDARY OUTCOMES:
FGF21 profile | 6 months after blood drawn
  FGF21 profile in first trimester of pregnancy and efficacy for GDM prediction

CONTACTS AND LOCATIONS:
Locations (1):
- Maharaj Nakorn ChiangMai Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided